CLINICAL TRIAL: NCT05477446
Title: Safety and Efficacy of CD207 Targeted CAR-T Cell Therapy in Patients With Relapsed and Refractory (R/R) Langerhans Cell Histiocytosis
Brief Title: Safety and Efficacy of CD207 Targeted CAR-T Cell Therapy in Patients With R/R Langerhans Cell Histiocytosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Boren Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Head of hematology, Principal Investigator, Clinical Professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRYY-IIT-LCYJ-2022-002
Record Dates: First submitted 2022-07-18; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: CAR-T cell therapy; Langerhans Cell histiocytosis; CD207
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD207 CAR-T cells (Experimental): Cohort 1 will receive 1 x 10^6 CAR+ T cells/kg. Cohort 2 will receive 3 x 10^6 CAR+ T cells/kg. Cohort 3 will receive 5 x 10^6 CAR+ T cells/kg. Cohort 4 will receive 1 x 10^7 CAR+ T cells/kg.
  Interventions: Biological: CD207 CAR-T cells

INTERVENTIONS:
Biological: CD207 CAR-T cells — Single dose of CD207 CAR-T cells administered IV

SUMMARY:
This is a single-arm study to evaluate the efficacy and safety of CD207 targeted CAR-T cell therapy in relapsed and refractory langerhans cell histiocytosis.

DETAILED DESCRIPTION:
There are limited options for treatment of r/r langerhans cell histiocytosis. CD207 is expressed on the membrane surface of langerhans cells，and it is an ideal target for CAR-T. In this study, investigators will evaluate the safety and efficacy of CD207 targeted CAR- T cell therapy in patients with r/r langerhans cell histiocytosis. The primary goal is safety and efficiency assessment, including incidence and severity of adverse events and overall response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory langerhans cell histiocytosis, defined as: 1) any relapse during standard chemotherapy; 2) not responding to standard chemotherapy; 3) not achieving CR after first cycle of second-line chemotherapy for relapsed langerhans cell histiocytosis;
2. 3-65 years old;
3. Expected survival time ≥ 3 months;
4. ECOG performance status of 0 or 1 (age ≥ 16 years) or Karnofsky performance status> 80 (age < 16 years) ;
5. With single or venous blood collection standards, and no other cell collection contraindications;
6. WBC ≥ 2.5×10^9/L ，LY ≥ 0.7×10^9/L，LY% ≥15%;
7. Serum creatinine ≤ 2.0 mg/dl;
8. ALT/AST ≤ 2.5 x ULN;
9. Total bilirubin ≤ 2.0 mg/dl;
10. PT:INR<1.7, or PT is within 4s of the normal value;
11. Ability and willingness to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

1. Transduced CAR+ T lymphocytes<5%, or expansion <5 folds after stimulation with anti CD3/anti CD28 beads;
2. Pregnant or breasting-feeding women;
3. Active hepatitis B or hepatitis C infection;
4. Patients with HIV infection;
5. Uncontrolled active infection;
6. Use of systemic corticosteroid therapy;
7. Have received gene therapy, or any other CAR-T treatment;
8. Allergic to immunotherapy and related drugs;
9. History of heart disease requiring treatment, or poorly controlled hypertension;
10. Preceding and/or ongoing active ulcer or gastrointestinal bleeding;
11. Have received allogeneic hematopoietic stem cell transplantation, or eligible for allogeneic hematopoietic stem cell transplantation;
12. Severe central nervous system involvement;
13. Severe lung involvement;
14. Hyponatremia (serum sodium<125mmol/L);
15. Hypokalemia (Serum kalium<3.5mmol/L);
16. Those who need long-term anticoagulation treatment (warfarin or heparin);
17. Those who need long-term antiplatelet treatment (aspirin, dose>300mg/d; clopidogrel, dose>75mg/d);
18. Radiation therapy within 4 weeks prior to registration;
19. Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, congestive heart failure, unstable angina, cardiac arrhythmias, mental illness, and other diseases that in the opinion of the investigator would pose an unacceptable risk to the subject;
20. Have a history of severe allergy;
21. Current enrollment in another study;
22. Patients with other contraindications considered unsuitable for participation in this study (according to investigator's judgement).

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 2 years
  The number of cases with complete response (CR) and partial response (PR) after treatment as a percentage of the total cases.
Incidence and Severity of Adverse Events (AEs) | 2 years
  Treatment-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) of CD207 CAR-T cell therapy in patients with r/r langerhans cell histiocytosis | 2 years
  PFS will be assessed from the first CAR-T cell infusion to death from any cause or the first assessment of progression.
Overall Survival (OS) of CD207 CAR-T cell therapy in patients with r/r langerhans cell histiocytosis | 2 years
  OS will be assessed from the first CAR-T cell infusion to death from any cause.
Effects of CD207 CAR-T cells on human immune system | 2 years
  Dynamic changes of T cell subset and immune globulin.
Metabolism of CAR T-cells in vivo | 2 years
  Absorption, distribution and metabolism of CD207-CAR T cells in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: ZHAO Wang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No